CLINICAL TRIAL: NCT00680082
Title: Observational Usage Study of Statins in Primary Care in France
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Russel Esterline, AstraZeneca
Other Study IDs: NIS-CFR-CRE-2007/2
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: statins; rosuvastatin; cross sectional study; France; CV risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients to whom a statin was initiated or switched between 3 and 6 months before consultation

SUMMARY:
To describe the way statins are used in France in primary care, that is to determine patients profile (particularly CV risk factors), to determine the way statins are initiated by general practitioners, to evaluate aftercare and to assess patients treated by rosuvastatin

ELIGIBILITY:
Inclusion Criteria:

* Patients to whom a statin was initiated or switched between 3 and 6 months before consultation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients recruited by a GP, community sample
Sampling Method: Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Morand, Principal Investigator — Cegedim Strategic Data - Boulogne Billancourt - France; Jean Dallongeville, Study Chair — Institut Pasteur - Inserm U744 - Lille -France
Locations (25):
- China (25):
  - Research Site, Hefei, Anhui
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Xiamen, Guangdong
  - Research Site, Zhongshan, Guangdong
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Jinan, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Rui’an, Zhejiang
  - Research Site, Wenzhou, Zhejiang